CLINICAL TRIAL: NCT04431635
Title: Phase IB Dose De-escalation Study of the PI3k Alpha/Delta Inhibitor, Copanlisib Given in Combination With the Immunotherapeutic Agents, Nivolumab and Rituximab in Patients With Relapsed/Refractory Indolent Lymphoma.Big Ten Cancer Research Consortium BTCRC-LYM17-145
Brief Title: Dose De-escalation Study of the PI3k Alpha/Delta Inhibitor, Copanlisib Given in Combination With the Immunotherapeutic Agents, Nivolumab and Rituximab in Patients With Relapsed/Refractory Indolent Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of study funding
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry); University of Michigan (Other); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2019.097; BTCRC-LYM17-145 (Other: BTCRC); HUM00166647 (Other: University of Michigan)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Indolent Lymphoma
MeSH Terms: interventions — copanlisib; Nivolumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A: Copanlisib, Nivolumab & Rituximab (Experimental): Copanlisib IV: day 1, 8, 15 every 28 days Nivolumab IV: Cycle 1 days 1 and 15; then day 1 only Rituximab IV: Cycle 1 days 1, 8, 15, 22; then day 1 (C2-6); then Q2 cycles (8-12)
  Interventions: Drug: Copanlisib; Drug: Nivolumab; Drug: Rituximab

INTERVENTIONS:
Drug: Copanlisib — Copanlisib IV: day 1, 8, 15 every 28 days
Drug: Nivolumab — Nivolumab IV: Cycle 1 days 1 and 15; then day 1 only
Drug: Rituximab — Rituximab IV: Cycle 1 days 1, 8, 15, 22; then day 1 (C2-6); then Q2 cycles (8-12)

SUMMARY:
Patients with relapsed or refractory follicular or marginal zone lymphoma who have received at least one prior line of therapy will receive

* Copanlisib IV: day 1, 8, 15 every 28 days
* Nivolumab IV: Cycle 1 days 1 and 15; then day 1 only
* Rituximab IV: Cycle 1 days 1, 8, 15, 22; then day 1 (C2-6); then Q2 cycles (8-12)

DETAILED DESCRIPTION:
Patients with relapsed/refractory lymphoma generally have few if any curative options and demonstrate poor response rates to standard salvage therapies. Novel regimens utilizing molecular targets are needed to improve outcomes in this patient population. While studies evaluating single agent small-molecule inhibitors have demonstrated activity in this setting, combinations of these drugs are generally thought to be more efficacious due to targeting separate mechanisms of action and decreased chance of developing resistance. The PD-1/PD-L1 axis is a molecular target that has been demonstrated to be up-regulated in several tumors including malignant lymphoma. Several pre-clinical studies have demonstrated the importance of this axis on clinical outcomes of patients afflicted with low grade lymphoma including FL. Targeting this axis with specific inhibitors would appear to be a rationale way to improve outcomes in patients afflicted with these diseases. PI3K inhibitors in addition to inhibiting signaling, impart changes in the immune cells in the tumor microenvironment and would appear to be a logical candidate to explore in combination with immunotherapy. Based on these preliminary data, we believe that we have justification for proceeding with our proposed phase I study to combine the PD-1 inhibitor, nivolumab, with the PI3K inhibitor, copanlisib, and the CD20 antibody, rituximab, in patients with relapsed/refractory follicular and marginal zone lymphoma. This work has the potential to provide a novel strategy to improve upon the clinical response noted in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of informed consent.
* Diagnosis of relapsed or refractory indolent follicular or marginal zone lymphoma established by histologic assessment by a hematopathologist that has relapsed after at least one line of chemo-immunotherapy.

  * Immunohistochemistry of the biopsy or
  * Flow cytometry of the biopsy
* ECOG Performance Status ≤ 2
* Has an indication for treatment based on the presence of symptoms and/or GELF criteria as referenced in appendix A.
* Must have failed or not be a candidate for an autologous stem cell transplantation.
* Women of childbearing potential must be willing to use appropriate contraception (barrier and hormonal therapy) or abstain from heterosexual activity from the point of registration through at least 12 months after the last dose of study drugs.

  -- NOTE: Women of childbearing potential are those who have not been surgically sterilized, have not been free of menses for ≥ 1 year, or her sole male partner has had a vasectomy at least 6 months prior to screening.
* Male subjects capable of fathering a child who have a female partner of childbearing potential must agree to use appropriate method(s) of contraception or abstain from heterosexual activity starting with the first dose of study drug through 1 month after the last dose of the study drugs.
* Adequate organ function defined as

  * Hepatic:

    * Total Bilirubin ≤ 1.5 mg/dL
    * AST and ALT ≤ 2.5 x ULN.
  * Renal: Creatinine < 2.0 mg/dl or CrCL > 30 mL/minute
  * Bone marrow function:

    * ANC ≥ 1000/mm3 (500/mm3 if known bone marrow (BM) involvement)
    * Platelet ≥ 75,000/mm3 (or 50,000/mm3 if known BM involvement)
    * Hgb > 9 g/dL (transfusions allowed to meet this criterion)
* Adequate glycemic control as demonstrated by a baseline fasting blood sugar (BS) ≤ 150 mg/dL. If uncontrolled then patient must be referred to PCP or endocrinology for medical management. Patient may be enrolled if adequate control is obtained prior to day 1 of therapy.
* Adequate blood pressure (BP) control as demonstrated by a baseline BP of < 150/90. If uncontrolled then patient must be referred to PCP for medical management. Patient may be enrolled if adequate control is obtained prior to day 1 of therapy.
* Prior treatment is allowed if

  * at least 4 weeks must have elapsed since last chemotherapy and/or radiation and the patient has recovered to ≤ grade 1 toxicity from all treatment related events.
  * at least 3 months must have passed since radio-immunotherapy.
  * at least 3 months have passed since date of stem cell infusion (autograft) and patient has recovered to ≤ grade 1 toxicities related to this procedure.
* Prior treatment with a PD-1/PD-L1 and/or PI3K inhibitor is allowed unless patient prior treatment was discontinued for intolerance.

Exclusion Criteria:

* Pregnant or breastfeeding women. NOTE: Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to study registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: Breast milk cannot be stored for future use while the mother is being treated on study.
* Diagnosis of follicular grade 3b, post-transplant lymphoproliferative disorder (PTLD), or presence of histologic transformation.
* Subjects with LFT abnormalities at baseline (above values per inclusion criteria), history of cirrhotic liver morphology or alcoholic cirrhosis, subjects who use acetaminophen at doses in excess of 2 g every day and have evidence of compromised hepatic reserve.
* Primary or metastatic CNS disease prior to study enrollment
* Uncontrolled current illness, including, but not limited to ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, evidence of interstitial lung disease or active, noninfectious pneumonitis including symptomatic and/or pneumonitis requiring treatment and/or psychiatric illness or social situations that would limit compliance with study requirements.
* History of inflammatory bowel disease i.e. Crohn's disease, ulcerative colitis.
* HIV infection. NOTE: HIV testing is required.
* Active infection with Hepatitis B or C virus (defined as a positive Hepatitis B surface antigen/ positive Hepatitis C antibody or detectable viral load by PCR). Patients with positive antibody but negative viral loads will be eligible for study participation but will require appropriate prophylaxis.

NOTE: Hepatitis B and C testing are required.

* Screening rate-corrected (using Friderica's correction) QT interval (QTcF) must not be > 480 msec via a standard 12-lead ECG within 28 days prior to registration.
* Concomitant therapy in the last 4 weeks of any of the following: cytotoxic chemotherapy, immunosuppressive agents, other investigational therapies, or chronic use of systemic corticosteroids (doses ≤ 10 mg/day prednisone or equivalent are permitted).
* Active or prior documented autoimmune or inflammatory disorders within the past 3 years prior to study registration. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (eg. following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment.
* Known allergy or reaction to any component of either study drug formulation.
* Prior allogeneic stem cell transplant.
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment.
* HbA1c > 8.5% at Screening
* Patient that require treatment with agents that are CYP3A4 inhibitors or strong CYP3A4 inducers. Patients who are on agents that fall into this category must be off for at least two weeks prior to start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
MTD (Maximum Tolerated Dose) of copanlisib given in combination with nivolumab and rituximab | 28 days
  To estimate the MTD (Maximum Tolerated Dose) of copanlisib given in combination with nivolumab and rituximab
Complete Response rate of the combination of copanlisib, nivolumab, and rituximab given at the MTD. | 1 year
  To estimate the Complete Response (CR) rate of the combination of copanlisib, nivolumab, and rituximab given at the MTD as determined by Lyric criteria [Cheson 2016}

SECONDARY OUTCOMES:
Summarize Adverse Events | Up to two years
  Summarize all adverse events graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall Response | 1 year
  The rate of overall response, defined as either CR or PR within 1 year of initiation of therapy.
Duration of Response | Up to two years
  3. Duration of response, as calculated from the time of initial response (CR or PR, determined by Lyric criteria [Cheson 2016]) until disease progression or death due to any cause (whichever occurs first).
Progression Free Survival | Up to two years
  4. Progression free survival, as calculated from the first dose of the combination to the occurrence of definitive disease progression (as defined by Cheson 2016) or death from any cause, whichever comes first.
Time to Next Treatment | Up to two years
  Time to next treatment (TTNT) is defined as the time from end of primary treatment to institution of next therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin H Karimi, MD, Principal Investigator — The University of Michigan Rogel Cancer Center
Locations (5):
- United States (5):
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No